CLINICAL TRIAL: NCT05768542
Title: Vacular Structure, Function and Sympathetic Activity in Takotsubo Syndrome
Brief Title: Sympathetic and Vascular Function in Takotsubo Syndrome
Acronym: SAFT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SAFT
Record Dates: First submitted 2023-01-26; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2022-10

CONDITIONS: Takotsubo Cardiomyopathy
MeSH Terms: conditions — Takotsubo Cardiomyopathy | interventions — Metoprolol; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Control group for primary outcome
Who Masked: Participant, Outcomes Assessor
Masking Description: Intervention single blinded to participant. Intervention blinded to person analyzing the MSNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Takotsubo Control (Active Comparator): Patients with Takotsubo receiving betablockade
  Interventions: Drug: Metoprolol Injection
- Takotsubo Intervention (Placebo Comparator): Patients with Takotsubo receiving placebo
  Interventions: Drug: Saline
- Control (No Intervention): Control subjects

INTERVENTIONS:
Drug: Metoprolol Injection — If heart rate below 60, give 5 mg IV. If heart rate above 60, give 5 mg IV and repeat until heart rate below 65 or 20 mg given in total or systolic blood pressure below 110 mmHg.
  Arms: Takotsubo Control
Drug: Saline — 5 ml given IV
  Arms: Takotsubo Intervention

SUMMARY:
The primary objective of this prospective, observational study is to compare muscle sympathetic nerve activity at rest and during stress between female patients with Takotsubo syndrome and healthy, matched volunteers.

* Do Takotsubo patients have an increased sympathetic nerve activity compared to controls?
* Do Takotsubo patients have an exaggerated sympathetic nerve activity response to stress?
* Does the sympathetic nerve activity response to stress in Takotsubo change after receiving the beta blocking agent metoprolol?

Participants will be examined with muscle sympathetic nerve activity recording in the peroneal nerve at rest and during cold pressor test. After intravenous injection with beta blocking agent (metoprolol) or placebo (saline) in a 1:1 randomized fashion, muscle sympathetic nerve recording at rest and during stress will be repeated.

DETAILED DESCRIPTION:
Female Takotsubo patients included in the SAFT (sympathetic and vascular function in Takotsubo syndrome) study will be invited to undergo microneurography recording of muscle sympathetic nerve activity (MSNA) at rest and during stress one week to two month after study inclusion. Responses to stress with and without the commonly used betablocking agent metoprolol will be compares.

Microneurography will be performed in the morning after a light caffeine-free breakfast with the subject supine and awake. Any medication with a beta blocking agent will be discontinued 24 hours prior to examination. MSNA will be recorded by inserting a tungsten electrode into the sympathetic nerve fibres of the peroneal nerve, with simultaneous blood pressure and heart rate monitoring.

MSNA recording will then continue during stress induced by placing one of the subjects hand in ice-cold water for 90 seconds (cold pressor test).

After intravenous injection with beta blocking agent (metoprolol) or placebo (saline) in a 1:1 randomized fashion, MSNA recording at rest and during stress will be repeated.

Age- and gender-matched healthy volunteers will be recruited as controls and examined similarly with microneurography at rest and during stress.

MSNA recordings will be amplified, computerized and saved for further analyses. MSNA will be quantified as burst incidence (burst per 100 heartbeats), burst frequence (bursts per minute) and relative median burst amplitude (%). MSNA activity will be compared between Takotsubo patients and controls and before and after betablockade in Takotsubo patients.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Diagnosis of Takotsubo cardiomyopathy

For Controls:

* Matching age with Takotsubo patients
* Signed informed consent

Exclusion Criteria:

* Coronary anathomy precluding intracoronary investigations
* Severe obstructive pulmonary disease
* Kidney failure with estimated glomerular filtration rate < 30 ml/min/m2
* Active malignancy
* Pericarditis

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Resting MSNA | During 5 minutes rest
  Muscle sympathetic nerve activity during rest
MSNA increase during CPT | During the last 60 seconds of the CPT
  Muscle sympathetic nerve activity increase during cold pressor test

SECONDARY OUTCOMES:
MSNA increase during CPT after intervention | During the last 60 seconds of the CPT
  Muscle sympathetic nerve activity increase during cold pressor test after betablockade
Hemodynamic changes during CPT | During the last 60 seconds of the CPT
  Change in blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Jonas 9, MD, PhD, Principal Investigator — Danderyd University Hospital and karolinska Institutet

IPD SHARING:
Plan to Share IPD: No
Needs approval according to GDPR but PI positive to requests